CLINICAL TRIAL: NCT06251973
Title: A Phase II Study of agenT-797 (Invariant Natural Killer T Cells), Botensilimab, a Novel Fc-enhanced CTLA-4 Inhibitor, Plus Balstilimab (Anti-PD-1) With Ramucirumab and Paclitaxel for Patients With Previously Treated, Advanced Esophageal, Gastric, or Gastro-esophageal Junction Adenocarcinoma
Brief Title: A Study of agenT-797 in Combination With Botensilimab, Balstilimab, Ramucirumab, and Paclitaxel for People With Esophageal, Gastric, or Gastro-esophageal Junction Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-361
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Esophageal Carcinoma; Advanced Unresectable Gastric Adenocarcinoma; Metastatic Gastric Cancer; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Esophageal Cancer; Metastatic Esophageal Adenocarcinoma; Metastatic Gastric Adenocarcinoma; Metastatic Gastric Carcinoma; Unresectable Esophageal Cancer; Unresectable Esophageal Adenocarcinoma; Unresectable Gastric Carcinoma; Unresectable Gastric Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma
Keywords: Metastatic Esophageal Carcinoma; Advanced Unresectable Gastric Adenocarcinoma; Metastatic Gastric Cancer; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Esophageal Cancer; Metastatic Esophageal Adenocarcinoma; Metastatic Gastric Adenocarcinoma; Metastatic Gastric Carcinoma; Unresectable Esophageal Cancer; Unresectable Esophageal Adenocarcinoma; Unresectable Gastric Carcinoma; Unresectable Gastric Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma; 23-261; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — balstilimab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants diagnoses with Esophageal, Gastric, or Gastro-esophageal Junction Cancer (Experimental): Participants with measurable disease and with evaluable disease as defined by RECIST v1.1 will be enrolled on this study.
  Interventions: Biological: AgenT-797; Biological: Botensilimab; Drug: Balstilimab; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Biological: AgenT-797 — AgenT-797 is an investigational product, composed of allogeneic human unmodified iNKT cells, isolated from mononuclear cell aphaeresis units from healthy donors
Biological: Botensilimab — Botensilimab is a novel, human, Fc-engineered IgG1 anti-CTLA-4 antibody
Drug: Balstilimab — Botensilimab is supplied as a sterile, single-use solution for IV administration
Drug: Ramucirumab — Ramucirumab is a fully human anti-VEGFR2 monoclonal IgG1 antibody (IgG1) that binds with high affinity to the extracellular domain of VEGFR2. Ramucirumab is a part of standard of care treatment for advanced gastric cancer or GEJ adenocarcinoma, after prior treatment with fluoropyrimidine- or platinum-containing chemotherarapy.
Drug: Paclitaxel — Paclitaxel is widely used across multiple cancer types and is a part of standard of care treatment for advanced EG adenocarcinoma after prior treatment with fluoropyrimidine- or platinum-containing chemotherarapy.

SUMMARY:
Participants will receive study treatment with agenT-797, botensilimab, balstilimab, ramucirumab, and paclitaxel. When participants start each agent will depend on how their disease is affecting them.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or advanced unresectable adenocarcinoma of esophageal, gastric, or gastroesophageal junction
* Disease progression on one prior line of therapy for metastatic disease. Patients with previously untreated advanced unresectable or metastatic disease may be included if disease progressed or recurred during neoadjuvant or adjuvant therapy or within 6 months of completion of those treatments.
* Patients must have histologically or cytologically confirmed esophageal, gastric, or gastroesophageal junction adenocarcinoma
* Patients must have measurable or evaluable disease as defined by RECIST v1.1 criteria. Patients with evaluable disease must be eligible to begin with an induction cycle
* Age 18 years or older
* ECOG performance status 0 to 1
* Adequate organ function as defined in Table 2

Table 2. Organ function requirements for eligibility Hematological Absolute neutrophil count: ≥1000/mcL Platelets: ≥90,000/mcL Hemoglobin: ≥8 g/dL Renal Serum creatinine: ≤1.5X ULN Hepatic Serum total bilirubin: ≤1.5X ULN OR Direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5X ULN, except patients with Gilbert's disease (≤3X ULN) AST and ALT: ≤2.5X ULN Albumin: ≥3 mg/dL

Exclusion Criteria:

* Received prior therapy with ramucirumab at any time
* Received paclitaxel or docetaxel-based therapy within 6 month of study enrollment
* Had a prior grade >3 immune related adverse event due to anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA4 therapy at any time
* Diagnosis of immunodeficiency or receipt of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment. Replacement therapy (ie physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic immunosuppressive therapy and is allowed.
* History of gastrointestinal perforation or fistulae
* A known history of active Bacillus tuberculosis
* Known active central nervous system metastases and/or carcinomatous meningitis
* History of or any evidence of active, non-infectious, immune-mediated pneumonitis. Patients with radiation-induced pneumonitis who are asymptomatic are permitted on study.
* Peripheral neuropathy limiting ADLs
* A known history of human immunodeficiency virus (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with HBsAg reactive on entecavir may be eligible after consultation with hepatologist and study team.
* Received a live vaccine within 30 days of planned start of study therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 5 months after the last dose of trial treatment
* Unwilling to give written, informed consent, unwilling to participate, or unable to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | up to 2 years
  Determine the efficacy of agenT-797, botensilimab and balstilimab in combination with ramucirumab and paclitaxel as second-line therapy in patients with advanced unresectable or metastatic esophagogastric cancer, as measured by ORR (defined as the percentage of patients who achieve either an objective complete response [CR] + partial response [PR])

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org